CLINICAL TRIAL: NCT00729820
Title: The Influence of Personality on Two Aspects of Cognitive Performance: Processing Speed, and Accuracy.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: BeerYaakov Mental Health Center (Other Government)
Responsible Party: dr kertzman semion, Beer-Yaakov MHC
Other Study IDs: cognitive performance-221CTIL
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-06

CONDITIONS: Healthy
Keywords: PERSONALITY; COGNITIVE PERFORMANCE; the practical usefulness (validity) of processing speed, accuracy of performance and personality measures in predicting impulsive behavior

SUMMARY:
Recently, a lot of evidence for a relation between measures of cognitive performance and personality characteristics has been collected. The use of computer based latency measures is often used to study mental processes in cognitive, as well as, in personality research On the basis of these relationships we can ask a question that relates to the practical usefulness (validity) of processing speed, accuracy of performance and personality measures in predicting impulsive behavior.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at age - 20-50 years

Exclusion Criteria:

* History of psychiatric disorders, previous hospitalizations and psychopharmacological treatments
* History of alcohol and substance abuse

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1. Men and women at age - 20-50 years
  2. The following demographic and anamnesis' data should be readily available:
  Age, ethnicity, marital and educational status. History of physical disorders and pharmacological treatments.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-08